CLINICAL TRIAL: NCT01628146
Title: PHASE IV STUDY # 1162. Prospective Investigation of SUPRACOR Visual Outcomes of Presbyopic Hyperopic Patients With and Without Astigmatism
Brief Title: Prospective Investigation of SUPRACOR Visual Outcomes of Presbyopic Hyperopic Patients With and Without Astigmatism
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Technolas Perfect Vision GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1162
Record Dates: First submitted 2012-06-06; First posted 2012-06-26 (Estimated); Last update posted 2015-05-20 (Estimated); Status verified 2015-05

CONDITIONS: Hyperopic Presbyopia
Keywords: Presbyopia; hyperopia; Supracor; contrast sensitivity
MeSH Terms: conditions — Presbyopia; Hyperopia | interventions — Keratomileusis, Laser In Situ

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SUPRACOR LASIK treatment (Experimental): SUPRACOR LASIK treatment
  Interventions: Device: SUPRACOR LASIK treatment

INTERVENTIONS:
Device: SUPRACOR LASIK treatment — The SUPRACOR algorithm uses the subjective refraction of the eye to create a treatment for the distance vision correction.
  Other Names: LASIK

SUMMARY:
This phase IV study is an open, prospective, single-center, single-surgeon bilateral eye study to investigate the bilateral uncorrected intermediate visual acuity of presbyopic hyperopic patients, who have been treated with Presbyopia Algorithm SUPRACOR.

DETAILED DESCRIPTION:
The developed software algorithm SUPRACOR uses the subjective refraction of the eye to create a treatment for the distance vision correction. This part of the treatment does not show any difference to a regular LASIK treatment for hyperopic cases. In addition to the treatment for the distance vision an additional central ablation component will be added to address the near vision.

Excimer Laser Technolas® 217z100P, High Speed Session Management Software (KERACOR V5.0) and ZYOPTIX Cards as well as all the diagnostic devices that are used in the #1162 study are CE certified and are used for their standard purpose.

This study will be conducted at Mater Private Hospital (Eye Laser Department) by Professor Michael O'Keefe who would recruit up to 40 subjects according to the inclusion/exclusion criteria.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be at least 48 years old and not older than 65 years
2. Subjects must read, understand, and sign an Informed Consent Form (ICF).
3. Subjects must be willing and able to return for scheduled follow up examinations through 6 months after surgery.
4. Subjects must be willing to have both eyes treated with the laser during the same visit.
5. Manifest Refraction for both eyes:

   * Sphere: +0.75 D to +5.00 D
   * Cylinder: -2.0 D to 0.0 D
   * Spherical Equivalent: +0.75 D to +4.0 D
6. Subjects must have presbyopia as determined by an age-related need for optical aid (≥+1.50 D) for reading with their best distance correction
7. The proper SUPRACOR treatment for the patient must target the dominant eyes for distance at 0.0/ 0.25 dpt and the following eye for near at -0.5/-0.75. The delta between the targets must remain 0.5 dpt
8. Subjects who have be screened successfully for acceptance of the SUPRACOR simulation
9. Subjects who are contact lens wearers must have gas permeable (GP) lenses discontinued for at least 3 weeks and soft lenses discontinued for at least 1 week prior to the preoperative evaluation in the eye to be treated. Contact lens wearers who wear their contact lenses for any amount of time between the preoperative baseline examination and the operative visit must not be treated.
10. Corneal topography should be normal.
11. Subjects who are contact lens wearers must have 2 central keratometry readings and 2 manifest subjective refractions taken preoperatively at least one week apart. The refraction values must not differ by more than 0.50 D as defined by manifest refraction spherical equivalent (MRSE). The keratometry values must not differ from the previous values by more than 0.50D in either meridian.
12. High contrast, manifest, best spectacle-corrected decimal distance visual acuity (VA) measured with the phoropter must be correctable to at least 1.0 (Snellen20/20 or 6/6) in both eyes.
13. Mesopic pupil size measured with Zywave II WaveFront Aberrometer and the special Pupil-o-Meter function must be between 3.5mm and 6.5 mm

Exclusion Criteria:

1. Subjects for whom the combination of their baseline corneal thickness and the planned operative parameters for the LASIK procedure would result in less than 250 microns of remaining posterior corneal thickness below the flap postoperatively.
2. Subject for whom a flap thickness other than 100-120µm is planed
3. Eyes for which the baseline manifest subjective refraction exhibits a difference of greater than 0.75D in sphere power, or a difference of greater than 0.50D in cylinder power, or a difference in cylinder axis of more than 15 degrees compared to the baseline cycloplegic subjective refraction. For manifest cylinder of less than 0.75D, the difference in cylinder axis will not be taken into consideration.
4. Subjects for whom the preoperative assessment of the ocular topography indicates that one or both eyes are not suitable candidates for treatment based upon the suggested computer-simulated treatment plan.
5. Any subject who is going to be co-managed by an ophthalmologist or optometrist who is not approved as a Technolas Perfect Vision GmbH Excimer laser Investigator.
6. Subjects with anterior segment pathology, including dry eye syndrome and cataracts which in the Investigator's opinion, would interfere with best spectacle-corrected VA (BSCVA) or a successful treatment.
7. Subjects with evidence of retinal vascular disease.
8. Subjects with any residual, recurrent, or active ocular disease, or corneal abnormality that in the Investigator's opinion would interfere with BSCVA or a successful treatment.
9. Subjects with signs of keratoconus.
10. Subjects with unstable central keratometry readings with irregular mires.
11. Subjects who have undergone previous intraocular or corneal surgery of any kind, including any type of Excimer laser surgery for either refractive or therapeutic purposes.
12. Subjects who have a history of Herpes simplex or Herpes zoster keratitis.
13. Subjects who have a history of glaucoma or glaucoma suspect.
14. Subjects who are immunocompromised or carrying diagnosis of connective tissue disease, clinically significant atopic disease, diabetes, autoimmune diseases and other acute or chronic illnesses that will increase the risk to the subject or confound the outcomes of this study.
15. Subjects taking systemic medications likely to affect wound healing such as corticosteroids or antimetabolites.
16. Subjects who are known to be pregnant, lactating, or who plan to become pregnant during the course of the study.
17. Subjects with known sensitivity to medications used for standard LASIK.
18. Subjects participating in any other ophthalmic study during this study.
19. Subjects with an ocular muscle disorder including a strabismus or nystagmus, or other disorders affecting fixation.
20. Subjects at risk for angle closure.
21. Subjects who have Diabetics
22. Subjects who have Cataract
23. Subject who have Dry Eye syndrome as evaluated with the "Tear Break Up-Time (TBUT)" Within this study protocol a TBUT ≥7 seconds is acceptable.

    -

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2012-09; Primary Completion 2015-07 (Estimated); Study Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
High contrast intermediate visual acuity | The study endpoints will be calculated for the 6-Month follow-up examination.
  The percentage of treated patients with a binocular uncorrected high contrast intermediate VA of 20/32 (0.4) or better. This percentage should be equal or greater than 60%.

SECONDARY OUTCOMES:
Contrast sensitivity | The study endpoints will be calculated for the 3-Month and 6-Month follow-up examination. The defined study endpoints should be fulfilled at least for the final examination at 6-Month.
  For all treated patients the mean value of the binocular photopic contrast sensitivity (log) for the various spatial frequencies should not decrease more than 0.30.
Patient satisfaction | The study endpoints will be calculated for the 3-Month and 6-Month follow-up examination. The defined study endpoints should be fulfilled at least for the final examination at 6-Month.
  The percentage of satisfied patient post SUPRACOR treatment. This percentage should be equal or greater than 75%.

CONTACTS AND LOCATIONS:
Overall Officials: Michael O'Keefe, MB, BAO, BcH, Principal Investigator — Mater Private Hospital, Dublin
Locations (1):
- Mater Private Hospital, Eye Laser Department, Dublin, Ireland